CLINICAL TRIAL: NCT03439943
Title: Multicenter, Randomised, Placebo-controlled, Double Blinded, Parallel Arm Proof-of-concept Trial of Lixisenatide in Patients With Early Parkinson's Disease
Brief Title: Study to Evaluate the Effect of Lixisenatide in Patient With Parkinson's Disease
Acronym: LixiPark
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Cure Parkinson's (Other); Réseau NS-Park (Unknown); EUCLID Clinical Trial Platform (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/16/8912
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — lixisenatide; Administration, Intravesical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lixisenatide (Experimental): Lixisenatide (10μg/d for 14 days and then 20μg/d): once daily subcutaneous
  Interventions: Drug: Lixisenatide
- Placebo (Placebo Comparator): Placebo: once daily subcutaneous injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lixisenatide — Patients randomized in the Lixisenatide group will receive 10μg/day for 14 days and then 20μg/day administered by once-daily subcutaneous injections during 12 months. If patients are unable to tolerable the dose of 20μg/day, this dose can be reduced to 10μg/day
  Other Names: injection drug
  Arms: Lixisenatide
Drug: placebo — Patients randomized in the placebo group will receive the corresponding placebo administered subcutaneously (once daily subcutaneous injection).
  Other Names: placebo injection
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the effect of lixisenatide (20 μg/d), versus placebo, administered as add-on therapy with the usual antiparkinsonian treatment, on the progression of motor disability in patients with early PD in order to assess its potential "disease-modifying" effect.

DETAILED DESCRIPTION:
This study will be a French, multicenter parallel groups, 2-arm, randomized, placebo-controlled, double-blind, proof-of-concept (POC) phase II trial evaluating the effect of lixisenatide, in patients with early PD.

The treatment period will be followed by a wash-out period of 2 months.

JUSTIFICATION/CONTEXT Parkinson's disease (PD) is a common neurodegenerative disease. Currently available symptomatic treatments allow improving motor and to a lesser extent non-motor function in PD patients.

None of these treatments can slow down the underlining disease process and the relentless progression of motor and non-motor disability.

Several mechanisms including the aggregation of misfolded alphasynuclein, mitochondrial dysfunction, oxidative stress and neuroinflammation have been related to the pathogenesis of PD. Recent evidence further suggests the implication of cerebral insulin resistance in the neurodegenerative process, while glucagon-like peptide 1 receptor (GLP1-R) agonists that are approved for the treatment of type 2 diabetes have neuroprotective properties in animal models of PD (Aviles-Olmos et al., 2013a). Moreover, the results of a recent clinical pilot trial suggest that treatment with the GLP-1R agonist exenatide for 12 months improves motor function in patients with moderate PD . GLP1-R are widely expressed in the central nervous system and GLP1-R agonists such as liraglutide, lixisenatide and exenatide have measurable brain concentrations, which makes them suitable for treating brain disorders.

Lixisenatide is a well-tolerated GLP-1R agonist that can be administered once-daily (subcutaneous injection). It has demonstrated positive effects on learning and memory through an increase of hippocampal neurogenesis in preclinical models of obesity/diabetes. Furthermore, lixisenatide increases neurogenesis and decreases microglial activation in rodent models of Alzheimer's disease (APPswe/PS1ΔE9 mice and Aβ25-35 rats) (. At the same dose, lixisenatide showed higher effectiveness at activating brain GLP-1R than liraglutide and exenatide, and showed more effective neuroprotection in a variety of in-vitro models of neurodegeneration (WO2013/030409A1).

Thus, this randomized, double-blind, clinical trial now aim to evaluate the effects of lixisenatide, versus placebo, on both motor and non-motor PD symptoms in patients at an early stage of PD.

This study will involve centers of the French national Parkinson's disease and movement disorders research network (Ns-Park network).

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD according to UKPDSBB criteria (male or female).
* Patient with a Hoehn and Yahr Stage <3 in the ON condition.
* Patients aged from 40 to 75 years old.
* Early-stage PD patients: diagnosis of PD for less than 3 years, without dyskinesia and motor fluctuations.
* Patients treated with an "optimized" stable dopaminergic medication regimen (dopamine agonist and/or L-dopa and/or MAOB inhibitor) for at least 1 month before baseline.
* Patients expected to remain on stable doses of antiparkinsonian medications for at least the first 6 months of the study and preferably for the 12 months of follow-up.
* Patients (or caregiver) able to self-administer lixisenatide injection.
* Patients with health insurance.
* Patients who signed the written informed consent form.

Exclusion Criteria:

* Patients suffering from other parkinsonian syndromes other than PD.
* Patients expected not to be able to remain on stable doses of symptomatic antiparkinsonian medications for at least 6-month.
* Patients with a Body Mass Index < 18.5
* Patients suffering from type 1 or type 2 diabetes.
* Malnutrition as assessed clinically by the investigator or any sub-investigator and by Mini Nutritional Assessment Short Form (MNA-SF) score <12 (the judgement of the investigator prevails over questionnaire scores).
* Weight change of more than 5 kg in body weight during the last 3 months prior to screening.
* Known history of drug or alcohol abuse within 6 months prior to the time of screening.
* Patients with hyperthyroidism or uncontrolled hypothyroidism. Note: Patients diagnosed with hypothyroidism need to be on a stable thyroid replacement therapy for at least 6 weeks.
* Patients with severe depression according to DSM criteria.
* Patients with cognitive impairment (MoCA score <26).
* Severe gastrointestinal disease (e.g. gastroparesis).
* Patients previously exposed to a GLP-1 agonist.
* Patients with severely impaired renal function (estimated creatinine clearance <30ml/min).
* Patients with a medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C (assessed by medical history), primary biliary cirrhosis, or ongoing symptomatic gallbladder disease.
* Patients with any clinically significant ECG abnormality.
* Laboratory findings at the time of screening:

Amylase and/or lipase: >3 times the upper limit of the normal (ULN) laboratory range ALT or AST: >3 times ULN Total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome) Calcitonin: >20 pg/mL (5.9 pmol/L) Hemoglobin: <11 g/dL (male/female) and/or neutrophils <1,500/mm3 and/or platelets <100,000/mm3 Triglyceride (TG): >600 mg/dL (6.78 mmol/L). History of unexplained pancreatitis, chronic pancreatitis or pancreatectomy.

* Personal or immediate family history of medullary thyroid cancer or genetic conditions that predispose to medullary thyroid cancer (e.g. multiple endocrine neoplasia syndromes).
* Hyperlipidemia.
* Females who are pregnant, breast feeding or of child bearing age without effective contraception.
* Patients treated per os in the evening by drugs requiring a rapid action (at the discretion of the investigator).
* Participants who lack the capacity to give informed consent.
* Any medical or psychiatric condition which may compromise participation in the study or the safety, at the discretion of the investigator.
* Known abnormality on CT or MRI brain imaging that is considered likely to compromise compliance with any aspect of the trial.
* Prior intra-cerebral surgical intervention for PD.
* Participant under legal guardianship or incapacitation.
* Patients who are participating or have participated in another interventional clinical trial within 30 days prior to baseline.
* Previous enrolment in the present trial.
* Allergic reaction to the active substance or to any of the excipients of lixisenatide

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end-point (M12) in the MDS-UPDRS III motor (Movement Disorder Society-Unified Parkinson's disease rating scale) | 12 month
  The main objective of the study is to evaluate the effect of lixisenatide (20 μg/d), versus placebo, administered as add-on therapy with the usual antiparkinsonian treatment, on the progression of motor disability in patients with early PD in order to assess its potential "disease-modifying" effect.
  The primary endpoint of this study is the change from baseline to end-point (M12) in the MDS-UPDRS III motor examination score, evaluated in the best ON condition in patients with early Parkinson's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier. RASCOL, MD, PHD, Principal Investigator — University Hospital, Toulouse
Locations (20):
- France (20):
  - University Hospital of Amiens, Amiens
  - University Hospital of Besancon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Caen, Caen
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - Creteil- Henri Mondor Hospital, Créteil
  - University Hospital of Lille, Lille
  - University Hospital of Limoges, Limoges
  - University Hospital of Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - Pitié Salpêtrière Hospital, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

REFERENCES:
- [Result] Meissner WG, Remy P, Giordana C, Maltete D, Derkinderen P, Houeto JL, Anheim M, Benatru I, Boraud T, Brefel-Courbon C, Carriere N, Catala H, Colin O, Corvol JC, Damier P, Dellapina E, Devos D, Drapier S, Fabbri M, Ferrier V, Foubert-Samier A, Frismand-Kryloff S, Georget A, Germain C, Grimaldi S, Hardy C, Hopes L, Krystkowiak P, Laurens B, Lefaucheur R, Mariani LL, Marques A, Marse C, Ory-Magne F, Rigalleau V, Salhi H, Saubion A, Stott SRW, Thalamas C, Thiriez C, Tir M, Wyse RK, Benard A, Rascol O; LIXIPARK Study Group. Trial of Lixisenatide in Early Parkinson's Disease. N Engl J Med. 2024 Apr 4;390(13):1176-1185. doi: 10.1056/NEJMoa2312323. PMID 38598572